CLINICAL TRIAL: NCT01569750
Title: A Phase 1b Study Combining Ibrutinib With Rituximab, Cyclophosphamide, Doxorubicin, Vincristine, and Prednisone (R-CHOP) in Subjects With CD20-Positive B-Cell Non Hodgkin Lymphoma (NHL)
Brief Title: A Study Combining Ibrutinib With Rituximab, Cyclophosphamide, Doxorubicin, Vincristine, and Prednisone in Patients With CD20-Positive B-Cell Non Hodgkin Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR100844; PCI-32765DBL1002 (Other: Janssen Research & Development, LLC); 2012-000546-35 (EudraCT Number)
Record Dates: First submitted 2012-03-30; First posted 2012-04-03 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: CD20-positive B-cell Non-Hodgkin Lymphoma
Keywords: CD20-positive B-cell non-Hodgkin lymphoma; Diffuse large B-cell lymphoma; Mantle cell lymphoma; Follicular lymphoma; Ibrutinib; R-CHOP; Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell; Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (1):
- Ibrutinib (Experimental): Part 1 (Dose Escalation): Escalating doses of ibrutinib (starting on Day 3 for Cycle 1 and on Day 1 for subsequent cycles) administered once daily in with standard-of-care doses of R-CHOP (rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisone) until maximum tolerated dose is achieved.
  Part 2: Ibrutinib at the recommended Part 1 dose administered once daily with standard-of-care doses of R-CHOP.
  Interventions: Drug: Part 1, Cohort 1; Drug: Part 1, Cohort 2; Drug: Part 1, Cohort 3; Drug: Part 2, Cohort 1; Drug: Part 2, Cohort 2

INTERVENTIONS:
Drug: Part 1, Cohort 1 — Type=exact number, unit=mg, number=280, form=capsule, route=oral use. Escalating doses of ibrutinib (starting on Day 3 for Cycle 1 and on Day 1 for subsequent cycles) administered once daily in with standard-of-care doses of R-CHOP until maximum tolerated dose is achieved.
Drug: Part 1, Cohort 2 — Type=exact number, unit=mg, number=420, form=capsule, route=oral use. Escalating doses of ibrutinib (starting on Day 3 for Cycle 1 and on Day 1 for subsequent cycles) administered once daily in with standard-of-care doses of R-CHOP until maximum tolerated dose is achieved.
Drug: Part 1, Cohort 3 — Type=exact number, unit=mg, number=560, form=capsule, route=oral use. Escalating doses of ibrutinib (starting on Day 3 for Cycle 1 and on Day 1 for subsequent cycles) administered once daily in with standard-of-care doses of R-CHOP until maximum tolerated dose is achieved.
Drug: Part 2, Cohort 1 — Ibrutinib at the recommended Part 1 dose administered once daily with standard-of-care doses of R-CHOP in patients with newly diagnosed diffuse large B-cell lymphoma.
Drug: Part 2, Cohort 2 — Ibrutinib at the recommended Part 1 dose administered once daily with standard-of-care doses of R-CHOP in patients with newly diagnosed with B-cell non-Hodgkin lymphoma.

SUMMARY:
The purpose of this study is to identify if, and at what dose, ibrutinib may be administered with R-CHOP (rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisone) and to document responses of this combination in patients with newly diagnosed diffuse large B-cell lymphoma (DLBCL).

DETAILED DESCRIPTION:
This is an open-label (individuals will know the identity of study treatments), dose escalation study to establish the recommended dose of ibrutinib combined with standard R-CHOP (rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisone) in approximately 33 adults with CD20-positive B-cell non-Hodgkin lymphoma (NHL) for whom R-CHOP is an appropriate therapy. There will be 3 periods of the study: a pretreatment (screening) period of up to 28 days before enrollment; an open-label treatment period (up to 6 cycles of ibrutinib and R-CHOP; ending at the end-of-treatment visit); and a posttreatment follow-up period until the end of study (maximum of up to 1 year after the last patient has completed the end-of-treatment visit). There are 2 parts to the study (dose escalation [Part 1] and expansion [Part 2]). During the dose escalation period, the "3+3" design will be applied and approximately 18 patients with CD20 positive B cell NHL (diffuse large B-cell lymphoma [DLBCL], mantle cell lymphoma [MCL], and follicular lymphoma [FL]) may be enrolled. Patients will be assigned to cohorts of increasing oral daily doses of ibrutinib (280, 420, and 560 mg) administered in combination with R-CHOP. The maximum tolerated dose (MTD), assessed in Cycle 1 (dose-limiting toxicity [DLT] period), is defined as the highest dose of the combination regimen at which <=33% of patients experience DLT. Baseline and follow-up electrocardiograms will be performed throughout the study. A Study Evaluation Team will review all available data upon completion of the first cycle for all patients at each dose cohort to determine DLTs, if dose escalation is acceptable, and subsequently will determine the recommended Phase 2 dose. Once the recommended Phase 2 dose is determined, approximately 15 patients with newly diagnosed DLBCL will be entered into the expansion cohort at the dose level selected to further assess the safety, pharmacokinetics, pharmacodynamics, pharmacogenomics, and activity of the combination. Patients whose disease has not progressed at the end of Cycle 1 will continue to receive ibrutinib and R CHOP up to a maximum of 6 cycles. During the posttreatment follow-up period, long term safety, survival status, disease progression, and subsequent antilymphoma therapy will be collected. The study will end 1 year after the last patient has completed the end of treatment visit.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically-confirmed CD20-positive B-cell non Hodgkin lymphoma disease for whom R-CHOP (rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisone) is an appropriate therapy (diffuse large B-cell lymphoma, mantle cell lymphoma, or follicular lymphoma); for the expansion cohort, at least 1 cohort will only include patients with newly diagnosed diffuse large B-cell lymphoma
* Stage I AX (bulk defined as single lymph node mass >=10 cm in diameter) to Stage IV disease
* At least 1 measurable site of disease based on the Revised Response Criteria for Malignant Lymphoma
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2
* Adequate bone marrow, liver, and renal function

Exclusion Criteria:

* History of protocol-defined disallowed therapies
* Prior multidrug chemotherapy treatment for lymphoma
* History of stroke or intracranial hemorrhage within 6 months prior to the first dose of study drug
* Major surgery within 3 weeks before enrollment
* Known bleeding diatheses, platelet dysfunction disorders, or requires therapeutic anticoagulation
* Known lymphoma of the central nervous system
* Uncontrolled or severe cardiovascular disease including myocardial infarction within 6 months of enrollment, New York Heart Association Class III or IV heart failure, uncontrolled angina, pericardial disease, cardiac amyloidosis, clinically significant cardiac arrhythmia, or left ventricular ejection fraction outside of institutional limits
* Active systemic infection requiring treatment including hepatitis B and hepatitis C infection
* Documented or suspected human immunodeficiency virus infection
* Diagnosed or treated for a malignancy other than non-Hodgkin lymphoma except; adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, ductal carcinoma in situ of the breast, or other solid tumors curatively treated with no evidence of disease for >5 years
* Has any condition that, in the opinion of the investigator, would make study participation not be in the best interest (eg, compromise the well-being) of the patient or that could prevent, limit, or confound the protocol-specified assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2012-06-14 (Actual); Primary Completion 2014-09-04 (Actual); Study Completion 2014-09-04 (Actual)

PRIMARY OUTCOMES:
Part 1 maximum tolerated dose of ibrutinib | Up to Cycle 1, Day 21 in Part 1
  The Part 1 maximum tolerated dose (MTD) is the Part 2 recommended ibrutinib dose.

SECONDARY OUTCOMES:
The number of participants affected by a dose-limiting toxicity | Up to Cycle 6, Day 21 in Part 1
Number of participants with potential drug-drug interactions between ibrutinib and vincristine | Up to Cycle 6, Day 21 in Part 2
Overall response rate | Up to Cycle 6, Day 21 in Part 2
Duration of response | Up to Cycle 6, Day 21 in Part 2
Progression-free survival | Up to Cycle 6, Day 21 in Part 2
Mean plasma concentrations of ibrutinib | Up to Cycle 6, Day 21 in Part 2
Maximum observed plasma concentration of ibrutinib | Up to Cycle 6, Day 21 in Part 2
Time to reach the maximum plasma concentration of ibrutinib | Up to Cycle 6, Day 21 in Part 2
Area under the plasma concentration-time curve from time 0 to 24 hours of ibrutinib | Up to Cycle 6, Day 21 in Part 2
Elimination half-life associated with the terminal slope of the semilogarithmic drug concentration-time curve of ibrutinib | Up to Cycle 6, Day 21 in Part 2
Elimination half-life associated with the terminal slope of the semilogarithmic drug concentration-time curve of vincristine | Up to Cycle 6, Day 21 in Part 2
Partial area under the plasma concentration versus time curve of vincristine | Up to Cycle 6, Day 21 in Part 2
The number of participants with pharmacodynamic markers of ibrutinib in peripheral blood mononuclear cells | Up to Cycle 6, Day 21 in Part 2
The number of participants with biomarkers predictive of clinical response | Up to Cycle 6, Day 21 in Part 2
The number of participants affected by an adverse event | Up to 30 days after the last dose of study medication

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (7):
- United States (4):
  - New York, New York
  - Rochester, New York
  - Nashville, Tennessee
  - Houston, Texas
- France (3):
  - Lille
  - Paris
  - Vandœuvre-lès-Nancy

REFERENCES:
- [Derived] Younes A, Thieblemont C, Morschhauser F, Flinn I, Friedberg JW, Amorim S, Hivert B, Westin J, Vermeulen J, Bandyopadhyay N, de Vries R, Balasubramanian S, Hellemans P, Smit JW, Fourneau N, Oki Y. Combination of ibrutinib with rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisone (R-CHOP) for treatment-naive patients with CD20-positive B-cell non-Hodgkin lymphoma: a non-randomised, phase 1b study. Lancet Oncol. 2014 Aug;15(9):1019-26. doi: 10.1016/S1470-2045(14)70311-0. Epub 2014 Jul 17. PMID 25042202
- See also: A Phase 1b Study Combining Ibrutinib with Rituximab, Cyclophosphamide, Doxorubicin, Vincristine, and Prednisone (R-CHOP) in Subjects with CD20-Positive B-Cell Non-Hodgkin Lymphoma (NHL) — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_7051&studyid=3512&filename=20150818_PCI-32765DBL1002_CSR_StudyReport.pdf